CLINICAL TRIAL: NCT00811850
Title: Comparing Effects of Two Fixed Combinations Ophthalmic Solutions on Ocular Blood Flow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GMA-COM-08-009
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Results first posted 2012-08-01 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Timolol; Ophthalmic Solutions; Brimonidine Tartrate, Timolol Maleate Drug Combination; dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combigan® (Active Comparator): Combigan® (fixed combination of brimonidine tartrate 0.2%/timolol maleate 0.5% ophthalmic solution). One drop of study medication taken approximately 12 hours apart, dosed 2 times a day for a total of two weeks.
  Interventions: Drug: fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5% ophthalmic solution
- Cosopt® (Active Comparator): Cosopt® (fixed combination of dorzolamide hydrochloride - timolol maleate ophthalmic solution). One drop of study medication taken approximately 12 hours apart, dosed 2 times a day for a total of two weeks.
  Interventions: Drug: fixed combination of dorzolamide hydrochloride timolol maleate ophthalmic solution

INTERVENTIONS:
Drug: fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5% ophthalmic solution — 1 drop of study medication taken approximately 12 hours apart, dosed 2 times a day for a total of two weeks
  Other Names: Combigan®
  Arms: Combigan®
Drug: fixed combination of dorzolamide hydrochloride timolol maleate ophthalmic solution — 1 drop of study medication taken approximately 12 hours apart, dosed 2 times a day for a total of two weeks
  Other Names: Cosopt®
  Arms: Cosopt®

SUMMARY:
A 10 week evaluation, crossover design study including a 3 week washout period between treatments, to determine the effects of Combigan® (fixed combination brimonidine tartrate 0.2%/timolol maleate 0.5%) and Cosopt® (fixed combination dorzolamide hydrochloride-timolol maleate ophthalmic solutions) on ocular blood flow as measured by retrobulbar blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30 years or older.
2. Primary open-angle glaucoma (POAG) or ocular hypertensive in at least one eye.
3. Best corrected visual acuity at least 20/40 in at least one eye.

Exclusion Criteria:

1. History of acute angle-closure or a narrow, occludable anterior chamber angle by gonioscopy.
2. History of chronic or recurrent inflammatory eye diseases (e.g., scleritis, uveitis).
3. History or signs of intraocular trauma.
4. Any abnormality preventing reliable applanation tonometry.
5. Current use of any ophthalmic or systemic steroid which may interfere with this investigation.
6. Severe, unstable or uncontrolled cardiovascular, renal, or pulmonary disease.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Indianapolis, Indiana, United States

REFERENCES:
- [Background] Siesky B, Harris A, Ehrlich R, Cantor L, Shoja MM, Rusia D, Hollander DA, Abrams L, Williams JM, Shoshani Y. Short-term effects of brimonidine/timolol and dorzolamide/timolol on ocular perfusion pressure and blood flow in glaucoma. Adv Ther. 2012 Jan;29(1):53-63. doi: 10.1007/s12325-011-0092-3. Epub 2012 Jan 11. PMID 22246943

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: This was a cross-over study with 3 treatment periods. In Treatment Period 1, patients received either Combigan® or Cosopt®. In Treatment Period 2, patients were washed out of their previous treatment. In Treatment Period 3, patients received either Combigan® or Cosopt® (treatment not received in Treatment Period 1).
Period: Treatment Period 1: Combigan® or Cosopt®
Arm/Group | All Patients
Started | 15
Completed | 15
Not Completed | 0
Period: Treatment Period 2: Wash Out
Arm/Group | All Patients
Started | 15
Completed | 15
Not Completed | 0
Period: Treatment Period 3: Combigan® or Cosopt®
Arm/Group | All Patients
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients in the study
Arm/Group | All Patients
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (NA) — Simple mean (average) was calculated for age. Standard deviation was not calculated. No other measure of dispersion was calculated.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Retrobulbar Blood Flow (Peak Systolic Velocity) as Measured by Color Doppler Imaging in the Nasal Short Posterior Ciliary Artery
Description: Peak systolic velocity (PSV) of retrobulbar blood flow as measured by color Doppler imaging (CDI) in the nasal short posterior ciliary artery after 1 month of treatment. CDI is a high-resolution ultrasound system which provides visualization of the flow of blood through a vessel. PSV is the maximum blood flow speed within a vessel at the time of systole (maximum pressure exerted in a blood vessel).
Time Frame: 1 Month
Population: Intent-to-treat population, which consisted of all patients that started the study (randomized)
Measure: Mean (Standard Deviation); unit: Centimeters per second (cm/s)
Arm/Group | Combigan® | Cosopt®
Number analyzed (Participants) | 15 | 15
Centimeters per second (cm/s) | 8.61 (2.33) | 8.02 (2.51)

2. Primary Outcome: Retrobulbar Blood Flow (End Diastolic Velocity) as Measured by Color Doppler Imaging in the Nasal Short Posterior Ciliary Artery
Description: End diastolic velocity (EDV) of retrobulbar blood flow as measured by color Doppler imaging (CDI) in the nasal short posterior ciliary artery after 1 month of treatment. CDI is a high-resolution ultrasound system which provides visualization of the flow of blood through a vessel. EDV is the maximum blood flow speed within a vessel at the end of diastole (minimum pressure exerted in a blood vessel in between heart beats).
Time Frame: 1 Month
Population: Intent-to-treat population, which consisted of all patients that started the study (randomized)
Measure: Mean (Standard Deviation); unit: Centimeters per second (cm/s)
Arm/Group | Combigan® | Cosopt®
Number analyzed (Participants) | 15 | 15
Centimeters per second (cm/s) | 2.63 (0.71) | 2.61 (0.63)

3. Primary Outcome: Retrobulbar Blood Flow (Peak Systolic Velocity) as Measured by Color Doppler Imaging in the Temporal Short Posterior Ciliary Artery
Description: Peak systolic velocity (PSV) of retrobulbar blood as measured by color Doppler imaging (CDI) in the temporal short posterior ciliary artery after 1 month of treatment. CDI is a high-resolution ultrasound system which provides visualization of the flow of blood through a vessel. PSV is the maximum blood flow speed within a vessel at the time of systole (maximum pressure exerted in the blood vessel).
Time Frame: 1 Month
Population: Intent-to-treat population, which consisted of all patients that started the study (randomized)
Measure: Mean (Standard Deviation); unit: Centimeters per second (cm/s)
Arm/Group | Combigan® | Cosopt®
Number analyzed (Participants) | 15 | 15
Centimeters per second (cm/s) | 8.52 (1.57) | 8.84 (1.75)

4. Primary Outcome: Retrobulbar Blood Flow (End Diastolic Velocity) as Measured by Color Doppler Imaging in the Temporal Short Posterior Ciliary Artery
Description: End diastolic velocity (EDV) of retrobulbar blood flow as measured by color Doppler imaging (CDI) in the temporal short posterior ciliary artery after 1 month of treatment. CDI is a high-resolution ultrasound system which provides visualization of the flow of blood through a vessel. EDV is the maximum blood flow speed within a vessel at the end of diastole (minimum pressure exerted in a blood vessel in between heart beats).
Time Frame: 1 Month
Population: Intent-to-treat population, which consisted of all patients that started the study (randomized)
Measure: Mean (Standard Deviation); unit: Centimeters per second (cm/s)
Arm/Group | Combigan® | Cosopt®
Number analyzed (Participants) | 15 | 15
Centimeters per second (cm/s) | 2.73 (0.67) | 2.87 (0.95)

5. Primary Outcome: Retrobulbar Blood Flow (Peak Systolic Velocity) as Measured by Color Doppler Imaging in the Ophthalmic Artery
Description: Peak systolic velocity (PSV) of retrobulbar blood flow as measured by color Doppler imaging (CDI) in the ophthalmic artery after 1 month of treatment. CDI is a high-resolution ultrasound system which provides visualization of the flow of blood through a vessel. PSV is the maximum blood flow speed within a vessel at the time of systole (maximum pressure exerted in a blood vessel).
Time Frame: 1 Month
Population: Intent-to-treat population, which consisted of all patients that started the study (randomized)
Measure: Mean (Standard Deviation); unit: Centimeters per second (cm/s)
Arm/Group | Combigan® | Cosopt®
Number analyzed (Participants) | 15 | 15
Centimeters per second (cm/s) | 24.5 (11.25) | 22.09 (8.25)

6. Primary Outcome: Retrobulbar Blood Flow (End Diastolic Velocity) as Measured by Color Doppler Imaging in the Ophthalmic Artery
Description: End diastolic velocity (EDV) of retrobulbar blood flow as measured by color Doppler imaging (CDI) in the ophthalmic artery after 1 month of treatment. CDI is a high-resolution ultrasound system which provides visualization of the flow through a vessel. EDV is the maximum blood flow speed within a vessel at the end of diastole (minimum pressure exerted in a blood vessel in between heart beats).
Time Frame: 1 Month
Population: Intent-to-treat population, which consisted of all patients that started the study (randomized)
Measure: Mean (Standard Deviation); unit: Centimeters per second (cm/s)
Arm/Group | Combigan® | Cosopt®
Number analyzed (Participants) | 15 | 15
Centimeters per second (cm/s) | 5.83 (2.49) | 5.18 (2.33)

7. Primary Outcome: Retrobulbar Blood Flow (Peak Systolic Velocity) as Measured by Color Doppler Imaging in the Central Retinal Artery
Description: Peak systolic velocity (PSV) of retrobulbar blood flow as measured by color Doppler imaging (CDI) in the central retinal artery after 1 month of treatment. CDI is a high-resolution ultrasound system which provides visualization of the flow of blood through a vessel. PSV is the maximum blood flow speed within a vessel at the time of systole (maximum pressure exerted in a blood vessel).
Time Frame: 1 Month
Population: Intent-to-treat population, which consisted of all patients that started the study (randomized)
Measure: Mean (Standard Deviation); unit: Centimeters per second (cm/s)
Arm/Group | Combigan® | Cosopt®
Number analyzed (Participants) | 15 | 15
Centimeters per second (cm/s) | 8.86 (2.19) | 8.81 (2.54)

8. Primary Outcome: Retrobulbar Blood Flow (End Diastolic Velocity) as Measured by Color Doppler Imaging in the Central Retinal Artery
Description: End diastolic velocity (EDV) of retrobulbar blood flow as measured by color Doppler imaging (CDI) in the central retinal artery after 1 month of treatment. CDI is a high-resolution ultrasound system which provides visualization of the flow of blood through a vessel. EDV is the maximum blood flow speed within a vessel at the end of diastole (minimum pressure exerted in a blood vessel in between heart beats).
Time Frame: 1 Month
Population: Intent-to-treat population, which consisted of all patients that started the study (randomized)
Measure: Mean (Standard Deviation); unit: Centimeters per second (cm/s)
Arm/Group | Combigan® | Cosopt®
Number analyzed (Participants) | 15 | 15
Centimeters per second (cm/s) | 2.73 (0.65) | 2.75 (0.78)

ADVERSE EVENTS:
Arm/Group | Combigan® | Cosopt®
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo